CLINICAL TRIAL: NCT06358703
Title: Impact of Acute ITTP Therapies on Long Term Neurologic and Cognitive Outcomes in ITTP Survivors
Acronym: NeST
Status: Not yet recruiting | Type: Observational
Sponsor: US Thrombotic Microangiopathy Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: P400
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-04

CONDITIONS: Immune Thrombotic Thrombocytopenia
Keywords: TTP; iTTP; aTTP; Cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — caplacizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma will be held in a biobank
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases
  Interventions: Drug: Caplacizumab
- Controls

INTERVENTIONS:
Drug: Caplacizumab — Early Caplacizumab use
  Groups: Cases

SUMMARY:
1. We expect to find that the silent cerebral infarct (SCI) rate is two fold higher in patients treated without caplacizumab. We also expect to find that the rate of mild and major cognitive impairment in patients treated with caplacizumab within 3 days of starting plasma exchange will be lower than patients treated without caplacizumab.
2. We expect that the differences in cognitive impairment in cases (caplacizumab) versus controls (no caplacizumab) will persist on serial evaluation 1 year later. We also expect that there will be differences in these groups even after adjusting for time since episode and severity of presentation.
3. We expect to find that SCI and cognitive impairment is associated with worse scores on the health related quality of life instrument (SF-36)
4. Based on studies in non-TTP populations, we expect to find that the rate of incident stroke over the period of follow up is at least 2 fold higher in patients that have SCI compared with patients who do not have SCI

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. Confirmed iTTP based on ADAMS13 activity < 10 % (or 10-20% with positive inhibitor or antibody) during an acute iTTP episode
3. Only 1 episode of iTTP that was treated with plasma exchange and caplacizumab started within 3 days of diagnosis (or if more than 1 episode, then all episodes treated with plasma exchange and caplacizumab started within 3 days of diagnosis)

Exclusion Criteria:

1. Any contraindication for MRI (metallic implants, shrapnel, MRI incompatible stents, etc)
2. Unable to speak, read or understand instructions in English (for NIH ToolBox)
3. Combination of iTTP episodes treated without caplacizumab or with caplacizumab.
4. Caplacizumab started at >= 4 days from diagnosis or for refractory iTTP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with iTTP
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Silent cerebral infarction | 12 months
  Silent cerebral infarction (primary endpoint) - SCI is derived from quantitation (number and total volume) of ischemic
  (infarct-like) lesions shown as foci of T2 and FLAIR hyperintensity. SCI is diagnosed if the participant has an infarct like
  lesion, at least 3 mm, with normal neurologic examination or an abnormality on examination that is not explained by the
  location of the brain lesion. We have assembled a panel of 3 neuroradiologists headed by Dr. Doris Lin. Each MRI will be
  read by 2 radiologists. A third reviewer will serve as a tie breaker in case of disagreement.
Cognitive impairment | 12 months
  Cognitive impairment (co-primary endpoint) - measured using NIH ToolBox Cognition Battery. Mild and major cognitive impairment are
  defined as T scores that are 1-2 SD below mean and > 2SD below mean for any domain, respectively

SECONDARY OUTCOMES:
Depression scores on BDI-II | 12 months
SF-36 scores for quality of life | 12 months
Patient reported cognitive performance | 12 months
  (PROMIS Cognitive Function - Short form 8a)

CONTACTS AND LOCATIONS:
Locations (1):
- USTMA, Groveport, Ohio, United States

IPD SHARING:
Plan to Share IPD: No